CLINICAL TRIAL: NCT06061016
Title: Construct Validity and Reliability of the 2-minute Step Test in Patients With Fibromyalgia
Brief Title: Validity and Reliability of the 2-minute Step Test in Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH2
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise test; Physical fitness
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of this study was twofold: first, to assess the validity and reliability of the 2 Minute Step Test (2MST) in patients with fibromyalgia; and second, to explore its relationship with objective assessment methods, specifically the 2 Minute Walk Test (2MWT) and the 6 Minute Walk Test (6MWT). Additionally, the study aimed to investigate the correlation between the 2MST and quality of life as well as chronic fatigue levels using the Fibromyalgia Impact Questionnaire (FIQ) and the Fatigue Severity Scale (FSS).

DETAILED DESCRIPTION:
This cross-sectional study will include 55 female patients aged 18-65 who will be diagnosed with fibromyalgia according to the American College of Rheumatology 2010 Diagnostic Criteria. Demographic characteristics of the patients will be documented. The extent of impact on patients' quality of life will be evaluated using the Fibromyalgia Impact Questionnaire (FIQ), while the severity of chronic fatigue will be measured using the Fatigue Severity Scale (FSS). The intensity of chronic pain experienced by patients will be expressed using the Visual Analogue Scale (VAS). All patients will undergo an initial assessment using the 2-Minute Step Test (2MST), 2-Minute Walk Test (2MWT), and 6-Minute Walk Test (6MWT). To assess test-retest reliability, the 2MST will be repeated with a 7-day interval between assessments.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with fibromyalgia according to the American College of Rheumatology 2010 Diagnostic Criteria
* Female patients aged 18-65
* The absence of any pathological condition that would hinder walking

Exclusion Criteria:

* Uncontrolled hypertension
* Decompensated heart failure
* Presence of systemic diseases affecting lower extremity functions
* Presence of degenerative diseases affecting lower extremity functions
* Peripheral artery disease causing vascular claudication
* Psychiatric illness
* Neuromuscular disease
* Pregnancy
* Cognitive impairment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Having been diagnosed with fibromyalgia according to the American College of Rheumatology 2010 Diagnostic Criteria
  * Female patients aged 18-65
  * The absence of any pathological condition that would hinder walking
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Two-minute step test | Baseline and Day 7
  The patient was instructed to lift their knees to the minimum marked level and take as many steps as possible in place for a duration of two minutes.

SECONDARY OUTCOMES:
Six-minute walk test | Baseline
  The distance the patient walked for six minutes was measured. An increase in the distance walked indicates improvement in basic mobility. The result is expressed in meters.
Two-minute walk test | Baseline
  The distance the patient walked for two minutes was measured. The result is expressed in meters.
Fibromyalgia Impact Questionaire | Baseline
  impact of life quality. The total score can be between 0-80 points. A score of 80 indicates maximum impact.
Fatigue Severity Scale | Baseline
  description fatigue level. The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on you. If 2.8<, no fatigue; If >6.1, chronic fatigue syndrome
Visual Analogue Scale | Baseline
  The pain VAS is a unidimensional measure of pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Kesiktas, MD, Study Chair — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCain A, McGibbon C, Carroll M, MacKenzie E, Senechal M, Bouchard DR. Validity of common physical function tests performed online for older adults. Arch Gerontol Geriatr. 2023 Nov;114:105104. doi: 10.1016/j.archger.2023.105104. Epub 2023 Jun 15. PMID 37354737
- [Background] de Morais Almeida TF, Dibai-Filho AV, de Freitas Thomaz F, Lima EAA, Cabido CET. Construct validity and reliability of the 2-minute step test in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2022 Feb 17;23(1):159. doi: 10.1186/s12891-022-05114-1. PMID 35177048
- [Background] de Jesus SFC, Bassi-Dibai D, Pontes-Silva A, da Silva de Araujo A, de Freitas Faria Silva S, Veneroso CE, de Paula Gomes CAF, Dibai-Filho AV. Construct validity and reliability of the 2-Minute Step Test (2MST) in individuals with low back pain. BMC Musculoskelet Disord. 2022 Dec 5;23(1):1062. doi: 10.1186/s12891-022-06050-w. PMID 36471309